CLINICAL TRIAL: NCT01607320
Title: Effect of Raloxifene on Ovulation in Women With Polycystic Ovarian Syndrome.
Brief Title: Efficacy Study of Raloxifene to Induce Ovulation in Polycystic Ovarian Syndrome
Acronym: PCOS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Over budget, slow recruitment, and personnel change
Sponsor: Bruce Lessey (Other)
Responsible Party: Sponsor-Investigator, Bruce Lessey, MD, PhD. and Professor of Clinical Obstetrics & Gynecology, Dept of OB/GYN, Prisma Health-Upstate
Organization: Prisma Health-Upstate (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9469
Record Dates: First submitted 2012-02-15; First posted 2012-05-30 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-08

CONDITIONS: Polycystic Ovarian Syndrome
Keywords: PCOS; Infertility; Anovulation
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility; Anovulation | interventions — Raloxifene Hydrochloride; Medroxyprogesterone Acetate; Clomiphene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raloxifene (Experimental): 3 cycles of 120mg/day of Evista (raloxifene) on days 3 to 7
  Interventions: Drug: Raloxifene
- Clomiphene (Active Comparator): 3 cycles of 100mg/day of Clomid (clomiphene citrate) on days 3 to 7
  Interventions: Drug: Clomiphene

INTERVENTIONS:
Drug: Raloxifene — Thirty PCOS patients treated with 3 cycles of 120mg/day of Evista (raloxifene) on days 3 to 7 following an initial provera withdrawal
  Other Names: Provera
  Arms: Raloxifene
Drug: Clomiphene — Thirty PCOS patients treated with 3 cycles of 100mg/day of Clomid (clomiphene citrate) on days 3 to 7 following an initial provera withdrawal
  Other Names: Provera
  Arms: Clomiphene

SUMMARY:
This study examines Raloxifene versus Clomiphene to induce ovulation in women with polycystic ovarian syndrome (PCOS).

DETAILED DESCRIPTION:
Clomiphene citrate (CC) is the major pharmaceutical treatment of anovulation in polycystic ovary syndrome, used for over 40 years. Despite the vast experience using this drug, the pregnancy rates associated with its use are low and recent large studies from Australia regarding birth defects suggest that CC may be associated with birth defects. Alternatives to CC are limited. Another selective estrogen receptor modulator, Raloxifene (RAL) does not have the long half life exhibited by CC, and has recently been shown to be equivalent to CC in terms of ability to induce ovulation in PCOS women. In addition, prior studies have demonstrated potential benefits on markers of uterine receptivity in a cell line model by blocking estrogen activity. Beyond this, there are no studies to examine whether Raloxifene is an effective oral agent for the treatment of women desiring pregnancy, but the investigators' hypothesis is that Raloxifene will work as well as CC but be better at establishment and maintenance of pregnancy than CC

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 to 36
2. BMI > 19 & < 40
3. PCOS diagnosis as evidenced by:

Oligo- and/or anovulation (< 6 cycles per year) and one of the following:

* Clinical and/or biochemical signs of hyperandrogenism
* Polycystic ovaries and exclusion of other aetiologies (congenital adrenal hyperplasias, androgen-secreting tumors, Cushing's syndrome)

Exclusion Criteria:

1. Use of ovulation induction agents within the past 6 months
2. Positive pregnancy test before taking study medications
3. History or current thromboembolic disorder
4. Coronary artery disease such as heart attack or stroke
5. Tobacco use or history within the past 6 months
6. History of pelvic inflammatory disease and tubal factor infertility
7. Congenital adrenal hyperplasia
8. Diabetes Mellitus

   * Any subject on Metformin must "wash out" for 30 days prior to screening
9. History of endometriosis
10. Known male factor infertility

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A. Lessey, MD, PhD, Principal Investigator — Greenville Hospital System
Locations (1):
- Greenville Hospital System, Greenville, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Raloxifene | Clomiphene
Started | 0 (The study was randomized between the two treatments and was never unblinded,therefore unknown.) | 0 (The study was randomized between the two treatments and was never unblinded,therefore unknown.)
Completed | 0 (The study was randomized between the 2 treatments and was never unblinded,so unknown.) | 0 (The study was randomized between the two treatments and was never unblinded,therefore unknown.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants were randomized to receive one of the two following interventions, but the study was terminated and data will not be unblinded: 1) 3 cycles of 120mg/day of Evista (raloxifene) on days 3 to 7 with Raloxifene: Thirty PCOS patients treated with 3 cycles of 120mg/day of Evista (raloxifene) on days 3 to 7 following an initial provera withdrawal; or 2) 3 cycles of 100mg/day of Clomid (clomiphene citrate) on days 3 to 7 with Clomiphene: Thirty PCOS patients treated with 3 cycles of 100mg/day of Clomid (clomiphene citrate) on days 3 to 7 following an initial provera withdrawal
Arm/Group | All Study Participants
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Pregnancy
Description: Time frame will vary depending on how many treatment cycles it takes to get pregnant. If no pregnancy occurs, study participation will likely be about 4 months.
Time Frame: 4 months
Population: The study was randomized between the two treatments and was never unblinded, therefore randomization is unknown and data collection is incomplete.
Groups:
- All Study Participants: The study was randomized between the two treatments and was never unblinded, threfore randomization is unknown.
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: Ovulation
Description: If ovulation does not occur during the first treatment cycle, subject will be withdrawn from study.
Time Frame: Cycle day 22-24
Population: Data collected could not be analyzed as it was never unblended and randomization is unknown.
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Study Participants (N=3)
headache (General disorders) | 1 — pt 3 experienced headace noted at visit 3
head cold (Infections and infestations) | 1 — pt 2 experienced head cold at visit 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No